CLINICAL TRIAL: NCT02123966
Title: An Open Label Phase II Trial of Topical Sirolimus for the Treatment of Refractory Oral Chronic Graft-versus-Host-Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow accrual, study team has decided to end the study early.
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Nathaniel S. Treister, DMD, DMSc, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-090
Record Dates: First submitted 2014-04-23; First posted 2014-04-28 (Estimated); Results first posted 2018-07-24 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-06

CONDITIONS: Chronic Graft-versus-Host-Disease; Oral Mucosal Disease Due to Graft-versus-host Disease
Keywords: Chronic Graft-versus-Host-Disease; Oral mucosal disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Topical Sirolimus + Steroid (Experimental): A four week supply of topical sirolimus will be dispensed. The treatment instructions will be to rinse and spit (NOT swallow) with one teaspoon (5 mL) of sirolimus solution 0.1mg/mL, combined with one teaspoon (5 mL) of steroid solution (dexamethasone 0.1%, clobetasol 0.05%, or budesonide 0.03%, based on the ongoing topical steroid prescription at the time of study enrollment) four times a day for 5 minutes at a time, and not to eat or drink for 15 minutes afterwards.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus
  Other Names: Rapamune®

SUMMARY:
This research study is evaluating the effectiveness of topical sirolimus combined with topical steroid therapy, as a possible treatment for oral cGVHD.

DETAILED DESCRIPTION:
Topical steroid therapy can be effective in managing oral cGVHD symptoms. However, a certain proportion of participants will not experience an adequate response to topical steroids and continue to have some degree of discomfort. Sirolimus is a non-steroidal immunosuppressive medication that has demonstrated efficacy in the management of cGVHD. Based on this, it is believed that a topical formulation applied inside the mouth may also demonstrate efficacy on a localized basis.

The purpose of this study is to assess the safety and efficacy of topical sirolimus as a swish and spit solution for the treatment of oral cGVHD in participants that have not had an adequate clinical response to topical steroid therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* While there will be no restrictions on concurrent systemic medications, all subjects must be on a stable immunomodulatory medication regimen for 7 days prior to beginning the study without plans to adjust doses during the following four-week study period. Dose modifications to maintain therapeutic drug levels of immunosuppressants (i.e. tacrolimus and sirolimus) during the study intervention period are allowed and do not constitute a trial violation. Changes in medications for non-cGVHD medical conditions will not affect eligibility.
* Age 4 years and older.
* Patients with symptomatic oral chronic graft-versus-host disease (sensitivity score ≥ 4).
* Stable topical steroid therapy with dexamethasone, clobetasol, or budesonide oral solutions (5 min, four times a day) for seven days prior to study enrollment.
* Stable systemic cGVHD medication regimen for seven days prior to study enrollment. Dose modifications to maintain therapeutic drug levels of immunosuppressants (i.e. tacrolimus and sirolimus) for the month prior and during the study intervention period are allowed and do not constitute a trial violation.
* The effects of sirolimus on the developing human fetus are unknown. For this reason and because immunosuppressants agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of topical sirolimus administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients already using topical sirolimus therapy.
* Patients who have an allergy/intolerance to sirolimus.
* Sensitivity score ≤ 3.
* Inability to comply with study instructions.
* Pregnant or breastfeeding.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded due to the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants, breastfeeding should be discontinued if the mother is treated with sirolimus.
* HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with sirolimus. In addition, these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel S Treister, DMD, DMSc, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jagasia MH, Greinix HT, Arora M, Williams KM, Wolff D, Cowen EW, Palmer J, Weisdorf D, Treister NS, Cheng GS, Kerr H, Stratton P, Duarte RF, McDonald GB, Inamoto Y, Vigorito A, Arai S, Datiles MB, Jacobsohn D, Heller T, Kitko CL, Mitchell SA, Martin PJ, Shulman H, Wu RS, Cutler CS, Vogelsang GB, Lee SJ, Pavletic SZ, Flowers ME. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: I. The 2014 Diagnosis and Staging Working Group report. Biol Blood Marrow Transplant. 2015 Mar;21(3):389-401.e1. doi: 10.1016/j.bbmt.2014.12.001. Epub 2014 Dec 18. PMID 25529383
- [Background] Slade GD. Derivation and validation of a short-form oral health impact profile. Community Dent Oral Epidemiol. 1997 Aug;25(4):284-90. doi: 10.1111/j.1600-0528.1997.tb00941.x. PMID 9332805

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from July 2014 to November 2016.
Period: Overall Study
Arm/Group | Topical Sirolimus + Steroid
Started | 10
Completed | 9
Not Completed | 1
Not completed — Intercurrent Illness | 1

BASELINE CHARACTERISTICS:
Population: The analysis population is comprised of all enrolled participants.
Arm/Group | Topical Sirolimus + Steroid
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 67 [41 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Subjective Sensitivity Score Response
Description: The sensitivity score is one question on a self-reported assessment tool from the NIH consensus documents. The question asks: "Your mouth sensitivity at its WORST" with a score 0-10, 10 being the worst. Response was defined as a 3 point reduction in sensitivity score from pre-to-post treatment.
Time Frame: Pre treatment and after the 28 day (4 weeks) cycle of treatment
Population: The analysis population is comprised of all treated participants.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Topical Sirolimus + Steroid
Number analyzed (Participants) | 10
percentage of participants | 20 [3.7 to 50.7]

2. Secondary Outcome: Change Pre-to-post Treatment in Oral Health Impact Profile Assessment
Description: Oral health related quality of life will be assessed before and after topical sirolimus therapy using the 14-item Oral Health Impact Profile instrument that measures subject's perceptions of the impact of oral conditions on their well-being.
Time Frame: Pre treatment and after the 28 day (4 weeks) cycle of treatment
Population: Data was not accessible and therefore the analysis was not conducted.
Arm/Group | Topical Sirolimus + Steroid
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were evaluated at the clinical exam at completion of protocol treatment, up to day 33.
Groups:
- Sirolimus: A four week supply of topical sirolimus will be dispensed. The treatment instructions will be to rinse and spit (NOT swallow) with one teaspoon (5 mL) of sirolimus solution 0.1mg/mL, combined with one teaspoon (5 mL) of steroid solution (dexamethasone 0.1%, clobetasol 0.05%, or budesonide 0.03%, based on the ongoing topical steroid prescription at the time of study enrollment) four times a day for 5 minutes at a time, and not to eat or drink for 15 minutes afterwards. Subjects will maintain a diary and record each dose, the length of time rinsing, and any adverse effects (e.g. transient burning).
  Sirolimus
Arm/Group | Sirolimus
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
This study was terminated early due to weak accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No